CLINICAL TRIAL: NCT02569281
Title: Effectiveness of the Inclusion of US-guided Percutaneous Electrolysis (EPE®) in Subacromial Pain Syndrome
Brief Title: US-guided Percutaneous Electrolysis (EPE®) in Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC 08-2015
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Pain
Keywords: Subacromial pain syndrome; Eccentric exercise; Pressure pain; US-guided percutaneous electrolysis
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- US-guided percutaneous electrolysis (Experimental): Patients will receive one weekly session for 5 weeks including best-evidence manual therapy and an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles. The exercise program will be asked to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 5 weeks. In addition, they will receive one session of US-guided percutaneous electrolysis. This intervention consists of the application of a galvanic electrical current with an acupuncture needle in the soft tissue, in this case the supraspinatus tendon.
  Interventions: Other: US-guided percutaneous electrolysis
- Eccentric exercise (Active Comparator): Patients will receive one weekly session for 5 weeks including best-evidence manual therapy and an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles. The exercise program will be asked to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 5 weeks.
  Interventions: Other: Eccentric exercise

INTERVENTIONS:
Other: US-guided percutaneous electrolysis — US-guided percutaneous electrolysis consists of the application of a galvanic electrical current with an acupuncture needle in the soft tissue, in this case the supraspinatus tendon.
  Arms: US-guided percutaneous electrolysis
Other: Eccentric exercise — An eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles will be learned by the patients allocated to this group
  Arms: Eccentric exercise

SUMMARY:
Scientific evidence of conservative management of subacromial pain syndrome is conflicting. There is evidence that eccentric exercise programs are effective at medium term for this pain condition. The inclusion of other therapeutic modalities is still controversial. A recent study suggests that the inclusion of US-guided percutaneous electrolysis combined with eccentric exercises can be effective at short-term for this condition. The objective of this randomized clinical trial is to determine the effectiveness at short- and long-term of the inclusion of US-guided percutaneous electrolysis (EPE®) into a eccentric exercise protocol for the management of patients with subacromial pain syndrome for pain, function, disability and pressure pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* unilateral shoulder complaints with duration of at least 3 months;
* an intensity of at least 4 on an 11-point numerical pain rating scale (NPRS) during arm elevation;
* a positive painful arc test during abduction
* at least one positive of the following tests: Hawkins-Kennedy test, Neer's sig, empty can test, drop arm or lift-off test

Exclusion Criteria:

* bilateral shoulder symptoms
* younger than 18 or older than 65 years
* history of shoulder fractures or dislocation
* cervical radiculopathy
* previous interventions with steroid injections
* fibromyalgia syndrome
* previous history of shoulder or neck surgery
* any type of intervention for the neck-shoulder area during the previous year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Changes in disability before and after the intervention | Baseline, one week after the last session, 3 months and 6 months after the last session
  The Disabilities of the Arm, Shoulder and Hand (DASH) will be used to determine the disability induced by shoulder pain

SECONDARY OUTCOMES:
Changes in pain intensity before and after the intervention | Baseline, one week after the last session, 3 months and 6 months after the last session
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area.
Changes in functionality before and after the intervention | Baseline, one week after the last session, 3 months and 6 months after the last session
  The Shoulder Pain and Disability Index (SPADI) questionnaire will be used to assess function of the uppr extremity related to shoulder pain
Changes in pressure pain sensitivity before and after the intervention | Baseline, one week after the last session, 3 months and 6 months after the last session
  Pressure pain thresholds will be assessed over the cervical spine, the hand, the deltoid muscle and the tibialis muscle
Self-perceived improvement | Baseline, one week after the last session, 3 months and 6 months after the last session
  A Global Rating of Change (GROC) from -7 (a very great deal worse) to +7 (a very great deal better) will be used to assess self-perceived improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] de Miguel Valtierra L, Salom Moreno J, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL. Ultrasound-Guided Application of Percutaneous Electrolysis as an Adjunct to Exercise and Manual Therapy for Subacromial Pain Syndrome: A Randomized Clinical Trial. J Pain. 2018 Oct;19(10):1201-1210. doi: 10.1016/j.jpain.2018.04.017. Epub 2018 May 16. PMID 29777953